CLINICAL TRIAL: NCT06600347
Title: Effect of DASH Diet and Progressive Muscle Relaxation on Cardiovascular Risks in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farahnaz Ahmed Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004059
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Complication
MeSH Terms: interventions — Dietary Approaches To Stop Hypertension; Autogenic Training; Antihypertensive Agents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DASH diet group (Experimental): The participants will be treated with the DASH diet and antihypertensive drugs
  Interventions: Dietary Supplement: DASH diet; Drug: Anti hypertensive drugs
- Progressive muscle relaxation group (Experimental): The participants will be treated with progressive muscle relaxation and antihypertensive drugs
  Interventions: Other: Progressive muscle relaxation; Drug: Anti hypertensive drugs
- DASH diet and progressive muscle relaxation group (Experimental): The participants will be treated with DASH diet and progressive muscle relaxation in addition to antihypertensive drugs
  Interventions: Dietary Supplement: DASH diet; Other: Progressive muscle relaxation; Drug: Anti hypertensive drugs

INTERVENTIONS:
Dietary Supplement: DASH diet — The participants will be treated with the DASH diet (1600-1800 calories/ day) for three months, in addition to antihypertensive drugs.
  Arms: DASH diet and progressive muscle relaxation group; DASH diet group
Other: Progressive muscle relaxation — The participants will be treated with progressive muscle relaxation for 30 minutes, 3 times/week for 3 months, in addition to antihypertensive drugs.
  Arms: DASH diet and progressive muscle relaxation group; Progressive muscle relaxation group
Drug: Anti hypertensive drugs — All participants in all groups will be treated with antihypertensive drugs as prescribed from the physician

SUMMARY:
This study will be conducted to investigate the effect of DASH diet and Progressive muscle relaxation on cardiovascular risks in postmenopausal women.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of morbidity and mortality in men and women, but the incidence of cardiovascular disease related deaths is higher in women than men. Hypertension is one of the leading risk factors for cardiovascular disease. Aging in both men and women is characterized by increases in blood pressure (BP), but the age-related increases are more rapid in women particularly postmenopausal women than in men.

A variety of non-pharmacologic treatments to manage stress have been found effective in reducing blood pressure and the development of hypertension. The DASH eating pattern promotes blood pressure reduction by encouraging the consumption of foods that are low in saturated fat, total fat, cholesterol, and sodium and high in potassium, calcium, magnesium, fiber, and protein. In terms of actual food choices, the DASH eating pattern encourages whole grains, fat free or low-fat dairy products, fruits, vegetables, poultry, fish, and nuts. Foods that are limited include fatty meats, full-fat dairy products, tropical oils (e.g., coconut, palm, and palm kernel oils), and sweets and sugar sweetened beverages.

The mechanism by which relaxation techniques lower blood pressure is unclear. One theory suggests that they may help lower the stress and physiologic arousal produced by the autonomic nervous system, thereby reducing blood pressure. So this study is a trial to determine the effect of DASH diet and progressive muscle relaxation in reducing cardiovascular risks in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* The participant's ages will be ranged from 50- 60 years old.
* Their body mass index will be ranged from 30-35 kg/m2.
* All women are hypertensive at least one year postmenopause.
* Their scores in perceived stress scale will be ranged from 14-40.

Exclusion Criteria:

* Women with systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) >100mmHg.
* Women who have other known causes of hypertension, such as renal diseases.
* Women who are using sedatives or tranquilizer or antidepressant drugs.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 3 months
  A sphygmomanometer will be used to measure systolic blood pressure (mmHg) for all participants in all groups before and after the treatment program
Diastolic blood pressure | 3 months
  A sphygmomanometer will be used to measure systolic blood pressure (mmHg) for all participants in all groups before and after the treatment program
Low density lipoprotein | 3 months
  Blood analysis will be used to measure level of low-density lipoprotein (mg/dl) for all participants in all groups before and after the treatment program. Its normal value is less than 100 mg/dl.
High density lipoprotein | 3 months
  Blood analysis will be used to measure level of high-density lipoprotein (mg/dl) for all participants in all groups before and after the treatment program. Its normal value is from 40 to more than 60 mg/dl.
Triglyceride level | 3 months
  Blood analysis will be used to measure the level of triglycerides (mg/dl) for all participants in all groups before and after the treatment program. Its normal value is less than 150 mg/dl.
Total cholesterol level | 3 months
  Blood analysis will be used to measure level of total cholesterol (mg/dl) for all participants in all groups before and after the treatment program. Its normal value is up to 200 mg/dl.

SECONDARY OUTCOMES:
Stress measurement | 3 months
  Perceived stress scale (PSS) will be used to assess the degree of stress for all participants in all groups before and after the treatment program.The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way.
  Scoring: PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 items scale can be made from questions 2, 4, 5 and 10 of the PSS 10 items scale. The higher the total score, the higher the perceived stress level.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Awad, professor, Study Director — Cairo University; Heba Abdel Halim, PHD, Study Director — National Institute of Nutrition; Hala Emara, professor, Study Chair — Cairo University
Locations (1):
- Farahnaz Ahmed Mohamed, Suez, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol